CLINICAL TRIAL: NCT02594111
Title: Anti-inflammatory Therapy During Percutaneous Coronary Intervention
Brief Title: Colchicine in Percutaneous Coronary Intervention
Acronym: Colchicine-PCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CARB-025-15S
Record Dates: First submitted 2015-10-30; First posted 2015-11-02 (Estimated); Results first posted 2020-07-10 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
Keywords: inflammation; percutaneous coronary intervention; coronary artery disease; colchicine
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Colchicine (Active Comparator): Colchicine 1.8 mg PO over 1 hour
  Interventions: Drug: Colchicine vs Placebo
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Colchicine vs Placebo

INTERVENTIONS:
Drug: Colchicine vs Placebo — Colchicine vs Placebo 1.8 mg PO over 1 hour

SUMMARY:
Inflammation in the arteries of the heart may increase the risk of cardiac death. The proposed research seeks to identify the potential beneficial role of a safe anti-inflammatory medication, colchicine, on reducing damage caused by opening up a blockage in the arteries of the heart. With its quick onset of action and excellent safety profile, colchicine may have the potential to reduce risk of major adverse events related to the heart. This research also seeks to better understand the role of neutrophils, the most common type of inflammatory white blood cell in the body, when there is damage to the heart.

DETAILED DESCRIPTION:
The investigators will use colchicine as a tool to elucidate the role of neutrophil activation during acute vascular injury, and to explore the association between neutrophil activation and adverse cardiovascular outcomes. Colchicine reduces cell surface expression of selections, adhesion molecules key to neutrophil recruitment after vascular injury. Daily colchicine use is associated with reduced adverse cardiovascular events in stable atherosclerosis. Using a clinical percutaneous coronary intervention (PCI) model, the investigators evaluate whether pre-procedural colchicine (1.8 mg oral load over one hour) reduces the rate of post-PCI adverse cardiovascular outcomes in the context of a double-blind placebo-controlled randomized study. The investigators will also characterize neutrophil biology in acute vascular injury and the effects of colchicine on neutrophil biology in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Referred for possible PCI

Exclusion Criteria:

* Colchicine use within 1 month
* History of colchicine intolerance
* Glomerular filtration rate <30mL/minute or on dialysis (due to the need to adjust colchicine dose in this setting)
* Active malignancy or infection (major confounder with increased inflammatory markers)
* History of myelodysplasia (due to suggested cautionary use of colchicine in this setting)
* High-dose statin load <24 hours prior to procedure (major confounder that is known to reduce inflammatory levels in 12 to 24 hours)
* Use of anti-inflammatory agents (except aspirin) within 5 halflives of the individual drug
* Use of strong Cytochrome P450, Family 3, Subfamily A, Polypeptide 4 (CYP3A4) and/or P-glycoprotein inhibitors (e.g. ritonavir, ketoconazole, clarithromycin, cyclosporine, diltiazem and verapamil, again due to drug interactions)
* Unable to consent
* Participating in a competing study
* Any significant condition or situation that may put the subject at higher risk, confound the study results or interfere with adherence to study procedures

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Actual)
Dates: Start 2013-05-30 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binita Shah, MD, Principal Investigator — Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY
Locations (1):
- Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Talmor N, Pillinger MH, Xia Y, Leonard A, Curovic F, Shah B. Neutrophil Activation and Adhesiveness in Coronary Artery Disease: Results From the COLCHICINE-PCI Biomarker Substudy. J Am Heart Assoc. 2024 Oct;13(19):e036701. doi: 10.1161/JAHA.124.036701. Epub 2024 Sep 30. PMID 39344637
- [Derived] Shah B, Pillinger M, Zhong H, Cronstein B, Xia Y, Lorin JD, Smilowitz NR, Feit F, Ratnapala N, Keller NM, Katz SD. Effects of Acute Colchicine Administration Prior to Percutaneous Coronary Intervention: COLCHICINE-PCI Randomized Trial. Circ Cardiovasc Interv. 2020 Apr;13(4):e008717. doi: 10.1161/CIRCINTERVENTIONS.119.008717. Epub 2020 Apr 16. PMID 32295417

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Colchicine | Placebo
Started | 366 | 348
Completed | 366 | 348
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colchicine | Placebo | Total
Number analyzed (Participants) | 366 | 348 | 714
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (9.7) | 65.8 (10.7) | 65.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 24 | 54
  Male | 336 | 324 | 660
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 75 | 79 | 154
  Not Hispanic or Latino | 291 | 269 | 560
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 19 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 85 | 75 | 160
  White | 268 | 253 | 521
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 366 | 348 | 714

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Peri-procedural Myocardial Necrosis
Description: troponin above the upper limit of normal (ULN)
Time Frame: 24 hours
Population: Although 714 patients had baseline measure, were randomized to colchicine or placebo, and underwent coronary angiography, but of these, 400 patients went on to stent placement and had primary outcome measured (as per protocol)
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 206 | 194
Participants | 118 | 122
Statistical Analysis 1: Comparison: Colchicine vs Placebo; Test type: Superiority; p < 0.05, Chi-squared

2. Secondary Outcome: Number of Participants With All-cause Mortality, Non-fatal MI, or Target Vessel Revascularization (TVR)
Description: all-cause mortality, non-fatal MI (universal definition), or target vessel revascularization (TVR)
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 206 | 194
Participants | 23 | 25

3. Secondary Outcome: Number of Participants With All-cause Mortality, Non-fatal MI, or TVR
Description: all-cause mortality, non-fatal MI (universal definition), or target vessel revascularization (TVR)
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 206 | 194
Participants | 35 | 36

4. Secondary Outcome: All-cause Mortality, Non-fatal MI, or TVR
Description: all-cause mortality, non-fatal MI (universal definition), or target vessel revascularization (TVR)
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 206 | 194
Participants | 48 | 48

5. Secondary Outcome: All-cause Mortality, Non-fatal MI, or TVR
Description: all-cause mortality, non-fatal MI (universal definition), or target vessel revascularization (TVR)
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 206 | 194
Participants | 57 | 57

6. Secondary Outcome: All-cause Mortality, Non-fatal MI, or TVR
Description: all-cause mortality, non-fatal MI (universal definition), or target vessel revascularization (TVR)
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 206 | 194
Participants | 65 | 63

7. Secondary Outcome: All-cause Mortality, Non-fatal MI, or TVR
Description: all-cause mortality, non-fatal MI (universal definition), or target vessel revascularization (TVR)
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 206 | 194
Participants | 67 | 67

8. Secondary Outcome: Number of Participants With Peri-procedural Myocardial Infarction (MI)
Description: SCAI definition
Time Frame: 24 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 206 | 194
Participants | 6 | 9

ADVERSE EVENTS:
Time Frame: For those who underwent diagnostic coronary angiogram only (n=314): 24 hours For those who underwent percutaneous coronary intervention (n=400), all AEs other than death, myocardial infarction, and target vessel revascularization: 30 days For those who underwent percutaneous coronary intervention (n=400), death, myocardial infarction, and target vessel revascularization: at least 2 years but up to 5 years
Description: Note that all AEs except for death, myocardial infarction, and target vessel revascularization were recorded for all patients (n=714), while death, myocardial infarction, and target vessel revascularization were only recorded for those undergoing percutaneous coronary intervention (n=400) and so the at risk numbers are different.
Arm/Group | Colchicine | Placebo
All-Cause Mortality (participants affected / at risk) | 26/206 | 29/194
Serious Adverse Events (participants affected / at risk) | 72/366 | 79/348
Other Adverse Events (participants affected / at risk) | 67/366 | 36/348
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Colchicine (N=366) | Placebo (N=348)
GI distress (Gastrointestinal disorders) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 2
Access site discomfort (Injury, poisoning and procedural complications) | 0 | 1
Hemodynamic instability (General disorders) | 0 | 2
Fever (Immune system disorders) | 0 | 2
Elevated creatinine (Renal and urinary disorders) | 1 | 2
Ischemic stroke (Vascular disorders) | 1 | 0
Fluid overload (General disorders) | 1 | 1
Bleeding (General disorders) | 0 | 2
all-cause mortality (Cardiac disorders) | 26/206 | 29/194
myocardial infarction (Cardiac disorders) | 18/206 | 19/194
target vessel revascularization (Cardiac disorders) | 16/206 | 14/194
PCI-related myocardial infarction (Cardiac disorders) | 23/206 | 23/194
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Colchicine (N=366) | Placebo (N=348)
Chest pain (Cardiac disorders) | 33 | 25 — Unrelated to study medication
Gastrointestinal symptoms (Gastrointestinal disorders) | 34 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT02594111/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT02594111/SAP_003.pdf